CLINICAL TRIAL: NCT06160648
Title: The Comparative Effectiveness of Mechanical Diagnosis and Therapy and Management According to the Cervical Spine Clinical Practice Guidelines in People With Neck Pain Who Exhibit Directional Preference: A Randomized Clinical Trial
Brief Title: The Comparative Effectiveness of Interventions in People With Neck Pain Who Exhibit Directional Preference
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Ronald Schenk, Clinical Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00002750
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Neck Pain
Keywords: Neck pain; Mechanical Diagnosis and Therapy; Clinical Practice Guidelines
MeSH Terms: conditions — Neck Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated to one of two treatment groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The primary investigator and the participants are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical Diagnosis and Therapy (MDT) (Experimental): MDT is a system of examination and intervention based on the patient's response to repeated end range neck movements.
  Interventions: Other: Management according to Mechanical Diagnosis and Therapy
- Cervical Spine Clinical Practice Guidelines (CPGs) (Active Comparator): The CPGs are guidelines for examination and intervention based on a summary of research conducted on people with neck pain.
  Interventions: Other: Management according to the Cervical Spine Clinical Practice Guidelines

INTERVENTIONS:
Other: Management according to Mechanical Diagnosis and Therapy — MDT management is based on the patient response to repeated end range movements.
  Arms: Mechanical Diagnosis and Therapy (MDT)
Other: Management according to the Cervical Spine Clinical Practice Guidelines — CPG management is based on clinical research regarding management of people with neck pain.
  Arms: Cervical Spine Clinical Practice Guidelines (CPGs)

SUMMARY:
The goal of this clinical trial is to compare physical therapy treatments in people with neck pain. The main aim is to compare the short-term effectiveness of physical therapy treatment for neck pain as delivered through Mechanical Diagnosis and Therapy (MDT) as compared to the Cervical Spine Clinical Practice Guidelines (CPGs) in patients with neck pain.

Participants will be randomly allocated to receive treatment according to MDT or CPG guidelines. Researchers will compare outcomes between the two groups over 1 year.

DETAILED DESCRIPTION:
Neck pain is one of the leading musculoskeletal causes of disability, second only to low back pain. A growing number of individuals with spine pathologies are seeking medical care; however, the overall increase in costs for spinal conditions is largely due to the growing cost per individual. The age-standardized rates of incidence, prevalence, and years lived with neck pain in North America are higher when compared globally. Due to these high rates and increases in medical care for individuals with spinal pathologies, further research is essential in developing the most efficacious treatment approach. Current evidence-based interventions to address musculoskeletal conditions of the neck are summarized in the 2017 revision of the Neck Pain Clinical Practice Guidelines (CPGs). The most recent revision includes 4 categories of neck pain: neck pain with mobility deficits, neck pain with headaches, neck pain with radiating pain, and neck pain with movement coordination impairment. These categories differ from the McKenzie Method of Mechanical Diagnosis and Therapy (known clinically as MDT) classifications of Derangement Syndrome, Dysfunction Syndrome, Postural Syndrome, and Spinal other Subgroups. Neck pain is one of the leading musculoskeletal causes of disability, second only to low back pain. A growing number of individuals with spine pathologies are seeking medical care; however, the overall increase in costs for spinal conditions is largely due to the growing cost per individual. The age-standardized rates of incidence, prevalence, and years lived with neck pain in North America are higher when compared globally. Due to these high rates and increases in medical care for individuals with spinal pathologies, further research is essential in developing the most efficacious treatment approach. Current evidence-based interventions to address musculoskeletal conditions of the neck are summarized in the 2017 revision of the Neck Pain Clinical Practice Guidelines (CPGs). The most recent revision includes 4 categories of neck pain: neck pain with mobility deficits, neck pain with headaches, neck pain with radiating pain, and neck pain with movement coordination impairment. These categories differ from the McKenzie Method of Mechanical Diagnosis and Therapy (known clinically as MDT) classifications of Derangement Syndrome, Dysfunction Syndrome, Postural Syndrome, and Spinal other Subgroups. The primary aim of this study is to compare outcomes in people treated according to MDT or the CPGs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are consecutively referred to physical therapy for the treatment of neck pain will be recruited from three hospital-based outpatient physical therapy clinics. Patients will be included if they demonstrate directional preference in the physical therapy initial examination.
2. Patients aged 18-90 years

Exclusion Criteria:

Patients will be excluded if they:

1. Have a history of spinal surgery
2. Have cervical instability, and/or vertebral basilar insufficiency
3. Have a serious medical condition such as cancer, spondylolisthesis, rheumatoid arthritis, ankylosing spondylitis, or other related autoimmune diseases
4. Are currently pregnant
5. Are positive for upper motor neuron signs
6. Are experiencing problems with dizziness, tinnitus, swallowing, or bowel and bladder dysfunction.
7. Do not experience directional preference in the physical therapy initial examination.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | 1 year
  The NDI is an outcome tool used to measure patient's perceived level of function in relation to their neck pain.

SECONDARY OUTCOMES:
Fear Avoidance Belief Questionnaire (FABQ) | 1 year
  The FABQ is an outcome tool used to measure a patient's fear in relation to their neck pain.
Numerical Pain Rating Scale (NPRS) | 1 year
  The NPRS is a tool used to measure the patient's perception of the neck pain on a scale ranging from 0-10 with 10 representing the worst pain possible.
Patient Specific Functional Scale (PSFS) | 1 year
  The PSFS is an outcome tool used to assess which particular functional activities are most impacted by their pain.
Global Rating of Change Scale (GROC) | 1 year
  The GROC is an outcome tool used independently to measure improvements in a patient's condition or as an anchor for other outcome measures.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Good Shepard Penn Partners, Radnor, Pennsylvania
  - WellSpan Health, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided